CLINICAL TRIAL: NCT05144100
Title: Primary Surgery Vs Primary Chemoradiation for Oropharyngeal Cancer (Scope Trial) - A Phase II/III Integrated Design Randomized Control Trial
Brief Title: Surgery Vs Chemoradiation for Oropharyngeal Cancer- A Phase II/III Integrated Design Randomized Control Trial
Acronym: SCOPE
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Collaborators: All India Institute of Medical Sciences (Other); Amrita Institute of Medical Sciences & Research Center (Other)
Responsible Party: Principal Investigator, Dr.Deepa Nair, Professor, Surgical Oncology, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3582
Record Dates: First submitted 2021-10-10; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma | interventions — Surgical Procedures, Operative; Neck Dissection; Endoscopy; Radiation; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: There will be two groups/arms in the study to evaluate the efficacy of primary surgery versus primary chemoradiation. Participants will be assigned to one of two or more groups for the duration of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Surgery +/- Neck Dissection (Experimental): Patients would undergo appropriate surgery via open, endoscopic, TLM, TORS or a combination. The primary and the neck would be addressed. For N0 neck, clearance of levels II-IV will be required, with levels I and/or V electively dissected at the discretion of the operating surgeon and based on extension of nodal disease. For N+ neck and tumors approaching to within 1cm of the midline, we recommend a contralateral neck dissection be performed as well of levels II-IV but to be done as per operating team's discretion. For lateralized lesions of the BOT and tonsil, ipsilateral neck dissection will be performed. A minimum of 18 lymph nodes per dissected side of the neck is required and will be subject to quality assurance review
  Interventions: Procedure: Surgery with or without Neck Dissection
- Arm 2 - Chemoradiation (Experimental): Patients will receive IMRT with normal tissue sparing techniques (70Gy/35# or 66Gy/ 30#) along with concurrent weekly cisplatin. Weekly cisplatin will be administered during IMRT at a dose of 40 mg/m2 IV on days 1, 8, 15, 22, 29, 36, and 43 for a total of up to 7 weekly doses, administered during the course of IMRT.
  For patients with T1-2 lateralized tonsil tumors with <1 cm invasion into the soft palate, no invasion of BOT, and N1 neck involvement, unilateral neck will be irradiated. The contralateral neck will be addressed for some BOT tumors<1cm or at the midline and may be considered in patients with N2 and N3status. For patients with residual neck disease after CCRT, a formal neck dissection will be performed. For patients with residual primary disease after CCRT, surgery for the primary will be performed if feasible.
  Interventions: Radiation: Radiation; Drug: Cisplatin based chemotherpay

INTERVENTIONS:
Procedure: Surgery with or without Neck Dissection — An appropriate surgery as open, endoscopic, TLM, TORS or a combination with or without neck dissection e.g. levels dissected, sparing or sacrifice of the SCM, accessory nerve, etc as per patient disease and status will be performed
  Other Names: appropriate surgery as open, endoscopic, TLM, TORS or a combination with or without neck dissection
  Arms: Arm 1 - Surgery +/- Neck Dissection
Radiation: Radiation — Patients will receive IMRT with normal tissue sparing techniques (70Gy/35# or 66Gy/ 30#) along with concurrent weekly cisplatin. Weekly cisplatin will be administered during IMRT at a dose of 40 mg/m2 IV on days 1, 8, 15, 22, 29, 36, and 43 for a total of upto 7 weekly doses, administered during the course of IMRT.
  Other Names: Radiotherapy with IMRT with normal tissue sparing techniques
  Arms: Arm 2 - Chemoradiation
Drug: Cisplatin based chemotherpay — Cisplatin (dose-40 mg/m2weekly,upto6-7cycles) cycle 1 will be administered within first 2 # of radiation. The rest of the cycles will be given weekly.
  Arms: Arm 2 - Chemoradiation

SUMMARY:
The oropharyngeal areas mainly comprises of the tonsil, base tongue (BOT), soft palate and the posterior pharyngeal wall. Traditionally, surgical resection of oropharyngeal cancers (OPC) was a standard procedure, often performed through mutilating incisions with mandibulotomies, rendering significant post-operative functional deficits. Over the past 2 decades, there has been a major shift in treatment strategy with a majority of these cancers now being treated by primary concurrent chemoradiation (CCRT) with a trend towards organ and function preservation.

DETAILED DESCRIPTION:
The oropharyngeal region primarily comprises the tonsil, base tongue (BOT), soft palate and posterior pharyngeal wall. Traditionally, surgical resection of oropharyngeal cancers (OPC) was a standard procedure, often performed through mutilating incisions with mandibulotomies, rendering significant post-operative functional deficits. Over the past 2 decades, there has been a major shift in treatment strategy with a majority of these cancers now being treated by primary concurrent chemoradiation (CCRT) with a trend towards organ and function preservation. The landmark trial determining effective treatment options for OPCs was by the RTOG group (0129) that provided strong evidence for HPV status being an independent prognostic factor for overall survival (OS) and progression-free survival (PFS), with these patients having significantly improved outcomes. Furthermore, after adjusting for demographics, T stage, N stage and smoking status, the HPV positive population had a 58% reduction in the risk of death and a 51% reduction in risk of progression or death. Most of the discussion today in HPV positive OPC is based on treatment- intensification to improve quality of life (QOL) measures.

A more concerning issue is the poor outcome, both survival, and QOL, seen in the "high-risk" HPV negative OPCs. When treated with radical CCRT, HPV negative patients have substantially reduced survival, both in terms of locoregional control (LRC) and OS. In the RTOG 0129, the HPV negative population had a 25.1% reduction in OS at 3 years (57.1% vs 82.4%) when compared to patients with HPV positive tumors. The locoregional relapse rate at 3 years was 21% higher in these patients (35.1% vs 13.6% for HPV positive tumors). Moreover, the salvage rates in oropharyngeal cancers that have undergone radical CCRT are quite low with only a third of the recurrences being amenable for salvage surgery. This led to a trend of intensification of management for these HPV negative tumors with altered fractionation schema,CCRT, multi-drug induction chemotherapy and targeted molecular therapies. Even with all these efforts, simply altering the method of radiation delivery, dosing and/or adding different types of concurrent chemotherapy is not seeming to be sufficient to improve oncologic outcomes in HPV negative tumors.

In the contemporary literature, an approach to further intensify treatment would be the addition of upfront surgery on this high-risk HPV negative OPCs. The recent advances in head neck surgery incorporate minimally invasive techniques and some focus around a transoral approach. These include transoral laser microsurgery (TLM) and transoral robotic surgery (TORS). Compared to the open approaches, these have minimal or no external incisions and do not require morbid access procedures. TLM is a surgical technique used in combination with an endoscope or direct laryngoscopy, operating microscope and a carbon dioxide (CO2) laser. TORS is performed using a robotic system, the arms of which are placed within the patient's mouth but controlled by a surgeon sitting at a remote console. The surgeon is provided with an endoscopically derived 3-dimensional view used to perform an enblocresection of the oropharyngeal tumor. Open surgery today incorporates modified techniques in osteotomy design, fixation and reconstruction methods to reduce and/or eliminate the traditional complications and have the additional advantage of direct visualization of the tumor. To add to this, radiotherapy techniques have also improved with more concentrated dosing obtained with intensity-modulated radiotherapy (IMRT) resulting in fewer complications.

Irrespective of the management received, patients with oropharyngeal tumors have a significant impact on the swallowing function and quality of life (QOL). Multiple factors are thought to contribute to the severity of this dysphagia, including multimodality therapy (surgery, RT, chemotherapy), total radiation dose, dosimetry to organs at risk (OAR) and intrinsic patient radiosensitivity and susceptibility to fibrosis. Majority of the current data on QOL are from single institution studies. Sinclair et al found that patients undergoing TORS for early OPCs have an initial decrease in mean dysphagia scores using the MD Anderson Dysphagia Inventory-Head and Neck (MDADI-HN) in the immediate postoperative period when compared to baseline pre-operative scores, although a gradual increasing improvement was observed over time. The global and physical subscales were most affected in the immediate postoperative period with the recovery of scores observed at last follow up. Postoperative chemotherapy predicted gastrostomy tube dependence for greater than 3 months. Hurtuk et al have shown a decrease from baseline immediately after surgery in speech, eating, aesthetic, social, and overall QOL domains, using the Head and Neck Cancer Inventory (HNCI). However, at 1 year, the health-related QOL in the aesthetic, social, and overall domains were high. Eating function and attitude were the only variables not returning to the high domain. In another population-based analysis of head neck cancers, oropharyngeal cancers had the second-highest prevalence of dysphagia, with 31% of patients demonstrating elevated episodes of aspiration relative to baseline greater than 1 year after receiving treatment. Weinstein et al reported long-term dependence on tracheostomy and gastrostomy was seen in 2.4% and 5%, respectively.(21) Even in the RTOG study,43% of the patients had severe long-term Grade 3 or 4 toxicity requiring a feeding tube/gastrostomy for more than 2 years or longer and death without cancer progression. Nichols et al recently attempted to answer some of these questions (ORATOR trial) in a randomized trial for early OPCs treated with CCRT versus TORS. They found the MDADI scores at 1-year were statistically superior in the RT arm (p = 0.042), but not meeting the definition of a clinically meaningful change (powered to detect a 10-point improvement). For the other QOL metrics, outcomes were similar at 1-year. Feeding tube rates were 3% in the RT arm vs 0% in the TORS arm. Even the rates of treatment-related grade ≥2 adverse events (AEs) were similar, with more neutropenia, constipation, and tinnitus in the RT arm and more trismus in the TORS arm. The findings of aspiration on modified barium swallow (MBS) have been significantly predictive of pneumonia in many trials of chemotherapy and IMRT in oropharyngeal cancer (p=0.017, Sensitivity 80%, Specificity 60%), and silent aspiration was evident on MBS studies in 63% of patients who developed pneumonia. In addition, pharyngeal residue in MBS studies was significantly associated with the development of pneumonia after chemotherapy and IMRT (p<0.01). These results offer compelling support for the examination of objective swallowing impairment (ie, "airway protection" and "pharyngeal transit") as these health-related endpoints cannot be obtained by patient-reported outcome (PROs) measures alone. Even the long-term results of RTOG 9111 study showed unknown mortality in 30% of the patients who received chemo-radiation, possibly due to silent aspiration. Hence, a lot of unanswered questions remain in determining the optimum management of OPCS that have minimal complications and maximum survival advantage.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology proven diagnosis of squamous cell carcinoma of the oropharynx, localized to the tonsil and/or lateralized tongue-base
2. ECOG Performance Status ≤2
3. Age ≥18 to 70 years
4. Anesthetic fitness obtained for surgery under general anesthesia
5. Resectable primary tumor with an anticipation of achieving resection free margins either by minimally invasive/open techniques
6. Clinical stage III or IV, i.e. T1-T2 or T3-T4 with N0-N3. Nodal disease withextranodal extension on clinical examination/imaging may be included at the surgeon's discretion, if the nodal disease is deemed resectable by the operating surgeon
7. HPV negative status determined by p16 status.
8. No distant metastases below the clavicles, based upon the following minimum diagnostic workup:

   1. History/physical examination by the physician.
   2. Imaging of the head and neck (Contrast enhanced MRI for local workup and Chest CT/PET-CT for distant metastatic workup)
9. Patients with no contraindications to Cisplatin chemotherapy and radiotherapy
10. Adequate organ function

    1. Hematological- Hb> 10 g/L, ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L.
    2. Liver functions- bilirubin ≤ 2 x upper limit normal (ULN), AST/ALT/ ALP ≤ 2.5 x ULN, S. albumin ≥ 30 g/L.
    3. Renal function- Creatinine ≤ 1.5 ULN, Creatinine clearance > 50 mL/min.
11. Women of child bearing age should have a negative pregnancy test at the time of randomization and should be willing to use adequate contraception during the treatment phase of the trial
12. Patients who can be followed up and must be able to provide informed consent prior to study entry

Exclusion Criteria:

1. Prior head and neck malignancy
2. Prior invasive malignancy, unless disease free for a minimum of 3 years
3. Prior chemotherapy for a different cancer administered within 3 years prior to registration
4. Patients who have received any neoadjuvant/ induction chemotherapy
5. Prior radiotherapy to the region of the head and neck that would result in overlap of radiation therapy fields
6. Unresectable primary or nodal disease involving the carotid vessels, prevertebral fascia or skull base
7. Large soft palate involvement >1 cm
8. Deep extension into larynx, pre-epiglottic space and deep invasion into extrinsic muscles of tongue
9. Calculated GFR < 50 cc/min
10. Patients who have uncontrolled cardiac comorbidity

    1. QTc prolongation (a value of >450 milliseconds)
    2. Ejection fraction below 50%
    3. Presence of regional wall akinesia
11. Presence of previous episode of thrombosis or embolism or presence of a prothrombotic condition in last 1 year
12. Presence of severe malnutrition as defined by body mass index of below 16kg per m2 or presence of weight loss of greater than 20% in last 6 months
13. Severe active co-morbidities such as severe cardiac failure, severe pulmonary compromise, type 1or 2 diabetes mellitus (Hb1ac of > 8 mg/dl) severe and active infections or life expectancy less than 6 months
14. Prior allergic reaction to cisplatin
15. Radiographic evidence of retropharyngeal and/or level VI metastasis
16. Patients on other investigational drugs within last 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 498 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival.(EFS) | 5 years after completion of last participant enrollment
  Event Free Survival will be defined as the time between the date of randomization till the date of recurrence of the disease (either local, regional or distant failure) or death due to disease.
Overall Survival (OS) | 5 years after completion of last participant enrollment
  Overall Survival (OS) will be defined as the time between the date of randomization and the date of death due any cause

SECONDARY OUTCOMES:
Disease free survival (DFS) | 5 years after completion of last participant enrollment
  Disease free survival (DFS) will be defined as the time between the date of randomization till the date of recurrence or second primary disease (either locoregional or distant).
Progression free survival (PFS) | 5 years after completion of last participant enrollment
  Progression of disease would be defined as an increase in any dimension of the disease or recurrence of disease
Locoregional control (LRC) | 5 years after completion of last participant enrollment
  Locoregional control (LRC) will be defined as the time between the date of randomization and the date of local or regional failure
Subjective Swallowing function | After 1 year (short term) and after 3 years(long term) from the date of enrollment
  evaluate the swallowing function using MBS with/without video assisted measure (Functional Endoscopic Evaluation of Swallo (FEES) or videofluroscopy)
M.D. Anderson Dysphagia Inventory Head and neck cancer-specific quality of life and patietn reproted outcomes (QOL and PROs) | After 1 year (short term) and after 3 years(long term) from the date of enrollment
  M.D. Anderson Dysphagia Inventory in the short-term after completion of 1year and long-term after completion of 3years post enrollment
EORTC HN35 Head and neck cancer-specific quality of life and patietn reproted outcomes (QOL and PROs) | After 1 year (short term) and after 3 years(long term) from the date of enrollment
  EORTC HN35 in the short-term after completion of 1year and long-term after completion of 3years post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Nair, MS(ENT),DNB, Principal Investigator — Tata Memorial Hospital, Mumbai, India
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
We will Decide to share once required permissions are obtained.

REFERENCES:
- [Result] Holsinger FC, Weber RS. Swing of the surgical pendulum: a return to surgery for treatment of head and neck cancer in the 21st century? Int J Radiat Oncol Biol Phys. 2007;69(2 Suppl):S129-31. doi: 10.1016/j.ijrobp.2007.05.044. PMID 17848281
- [Result] WARD GE, ROBBEN JO. A composite operation for radical neck dissection and removal of cancer of the mouth. Cancer. 1951 Jan;4(1):98-109. doi: 10.1002/1097-0142(195101)4:13.0.co;2-r. No abstract available. PMID 14801776
- [Result] Golusinski W, Golusinska-Kardach E. Current Role of Surgery in the Management of Oropharyngeal Cancer. Front Oncol. 2019 May 24;9:388. doi: 10.3389/fonc.2019.00388. eCollection 2019. PMID 31179239
- [Result] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Result] Adelstein DJ, Ismaila N, Ku JA, Burtness B, Swiecicki PL, Mell L, Beitler JJ, Gross N, Jones CU, Kaufman M, Le QT, Semrad TJ, Siu LL, Ridge JA. Role of Treatment Deintensification in the Management of p16+ Oropharyngeal Cancer: ASCO Provisional Clinical Opinion. J Clin Oncol. 2019 Jun 20;37(18):1578-1589. doi: 10.1200/JCO.19.00441. Epub 2019 Apr 25. PMID 31021656
- [Result] Kano S, Homma A, Hayashi R, Kawabata K, Yoshino K, Iwae S, Hasegawa Y, Nibu K, Kato T, Shiga K, Matsuura K, Monden N, Fujii M. Salvage surgery for recurrent oropharyngeal cancer after chemoradiotherapy. Int J Clin Oncol. 2013 Oct;18(5):817-23. doi: 10.1007/s10147-012-0449-x. Epub 2012 Jul 25. PMID 22829207
- [Result] Brizel DM, Albers ME, Fisher SR, Scher RL, Richtsmeier WJ, Hars V, George SL, Huang AT, Prosnitz LR. Hyperfractionated irradiation with or without concurrent chemotherapy for locally advanced head and neck cancer. N Engl J Med. 1998 Jun 18;338(25):1798-804. doi: 10.1056/NEJM199806183382503. PMID 9632446
- [Result] Forastiere AA, Goepfert H, Maor M, Pajak TF, Weber R, Morrison W, Glisson B, Trotti A, Ridge JA, Chao C, Peters G, Lee DJ, Leaf A, Ensley J, Cooper J. Concurrent chemotherapy and radiotherapy for organ preservation in advanced laryngeal cancer. N Engl J Med. 2003 Nov 27;349(22):2091-8. doi: 10.1056/NEJMoa031317. PMID 14645636
- [Result] Forastiere AA, Zhang Q, Weber RS, Maor MH, Goepfert H, Pajak TF, Morrison W, Glisson B, Trotti A, Ridge JA, Thorstad W, Wagner H, Ensley JF, Cooper JS. Long-term results of RTOG 91-11: a comparison of three nonsurgical treatment strategies to preserve the larynx in patients with locally advanced larynx cancer. J Clin Oncol. 2013 Mar 1;31(7):845-52. doi: 10.1200/JCO.2012.43.6097. Epub 2012 Nov 26. PMID 23182993
- [Result] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Result] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Result] Holsinger FC, Sweeney AD, Jantharapattana K, Salem A, Weber RS, Chung WY, Lewis CM, Grant DG. The emergence of endoscopic head and neck surgery. Curr Oncol Rep. 2010 May;12(3):216-22. doi: 10.1007/s11912-010-0097-0. PMID 20425082
- [Result] McGregor IA, MacDonald DG. Mandibular osteotomy in the surgical approach to the oral cavity. Head Neck Surg. 1983 May-Jun;5(5):457-62. doi: 10.1002/hed.2890050512. PMID 6874369
- [Result] Spiro RH, Gerold FP, Strong EW. Mandibular "swing" approach for oral and oropharyngeal tumors. Head Neck Surg. 1981 May-Jun;3(5):371-8. doi: 10.1002/hed.2890030505. PMID 6263826
- [Result] Singh AM, Bahadur S, Tandon DA, Pande RM. Anterior mandibulotomy for oral and oropharyngeal tumours. J Laryngol Otol. 1993 Apr;107(4):316-9. doi: 10.1017/s0022215100122911. PMID 8320517
- [Result] Roux M, Dassonville O, Ettaiche M, Poissonnet G, Sudaka A, Bozec A. Transoral-transcervical oropharyngectomy without mandibulotomy, associated to fasciocutaneous radial forearm free-flap reconstruction, for oropharyngeal cancer: Postoperative course, oncologic and functional results, and prognostic factors. Eur Ann Otorhinolaryngol Head Neck Dis. 2017 Apr;134(2):71-76. doi: 10.1016/j.anorl.2016.11.004. Epub 2016 Nov 30. PMID 27914910
- [Result] Na HY, Choi EJ, Choi EC, Kim HJ, Cha IH, Nam W. Modified mandibulotomy technique to reduce postoperative complications: 5-year results. Yonsei Med J. 2013 Sep;54(5):1248-52. doi: 10.3349/ymj.2013.54.5.1248. PMID 23918577
- [Result] Sinclair CF, McColloch NL, Carroll WR, Rosenthal EL, Desmond RA, Magnuson JS. Patient-perceived and objective functional outcomes following transoral robotic surgery for early oropharyngeal carcinoma. Arch Otolaryngol Head Neck Surg. 2011 Nov;137(11):1112-6. doi: 10.1001/archoto.2011.172. PMID 22106235
- [Result] Hurtuk AM, Marcinow A, Agrawal A, Old M, Teknos TN, Ozer E. Quality-of-life outcomes in transoral robotic surgery. Otolaryngol Head Neck Surg. 2012 Jan;146(1):68-73. doi: 10.1177/0194599811421298. Epub 2011 Aug 31. PMID 21881053
- [Result] Francis DO, Weymuller EA Jr, Parvathaneni U, Merati AL, Yueh B. Dysphagia, stricture, and pneumonia in head and neck cancer patients: does treatment modality matter? Ann Otol Rhinol Laryngol. 2010 Jun;119(6):391-7. doi: 10.1177/000348941011900605. PMID 20583737
- [Result] Weinstein GS, O'Malley BW Jr, Desai SC, Quon H. Transoral robotic surgery: does the ends justify the means? Curr Opin Otolaryngol Head Neck Surg. 2009 Apr;17(2):126-31. doi: 10.1097/MOO.0b013e32832924f5. PMID 19342953
- [Result] Nichols AC, Theurer J, Prisman E, Read N, Berthelet E, Tran E, Fung K, de Almeida JR, Bayley A, Goldstein DP, Hier M, Sultanem K, Richardson K, Mlynarek A, Krishnan S, Le H, Yoo J, MacNeil SD, Winquist E, Hammond JA, Venkatesan V, Kuruvilla S, Warner A, Mitchell S, Chen J, Corsten M, Johnson-Obaseki S, Eapen L, Odell M, Parker C, Wehrli B, Kwan K, Palma DA. Radiotherapy versus transoral robotic surgery and neck dissection for oropharyngeal squamous cell carcinoma (ORATOR): an open-label, phase 2, randomised trial. Lancet Oncol. 2019 Oct;20(10):1349-1359. doi: 10.1016/S1470-2045(19)30410-3. Epub 2019 Aug 12. PMID 31416685
- [Result] Eisbruch A, Lyden T, Bradford CR, Dawson LA, Haxer MJ, Miller AE, Teknos TN, Chepeha DB, Hogikyan ND, Terrell JE, Wolf GT. Objective assessment of swallowing dysfunction and aspiration after radiation concurrent with chemotherapy for head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):23-8. doi: 10.1016/s0360-3016(02)02712-8. PMID 12007937
- [Result] Hunter KU, Schipper M, Feng FY, Lyden T, Haxer M, Murdoch-Kinch CA, Cornwall B, Lee CS, Chepeha DB, Eisbruch A. Toxicities affecting quality of life after chemo-IMRT of oropharyngeal cancer: prospective study of patient-reported, observer-rated, and objective outcomes. Int J Radiat Oncol Biol Phys. 2013 Mar 15;85(4):935-40. doi: 10.1016/j.ijrobp.2012.08.030. Epub 2012 Oct 3. PMID 23040224
- [Result] de Almeida JR, Byrd JK, Wu R, Stucken CL, Duvvuri U, Goldstein DP, Miles BA, Teng MS, Gupta V, Genden EM. A systematic review of transoral robotic surgery and radiotherapy for early oropharynx cancer: a systematic review. Laryngoscope. 2014 Sep;124(9):2096-102. doi: 10.1002/lary.24712. Epub 2014 May 27. PMID 24729006
- [Result] Yeh DH, Tam S, Fung K, MacNeil SD, Yoo J, Winquist E, Palma DA, Nichols AC. Transoral robotic surgery vs. radiotherapy for management of oropharyngeal squamous cell carcinoma - A systematic review of the literature. Eur J Surg Oncol. 2015 Dec;41(12):1603-14. doi: 10.1016/j.ejso.2015.09.007. Epub 2015 Sep 26. PMID 26461255
- [Result] Housset M, Baillet F, Dessard-Diana B, Martin D, Miglianico L. A retrospective study of three treatment techniques for T1-T2 base of tongue lesions: surgery plus postoperative radiation, external radiation plus interstitial implantation and external radiation alone. Int J Radiat Oncol Biol Phys. 1987 Apr;13(4):511-6. doi: 10.1016/0360-3016(87)90065-4. PMID 3558042
- [Result] Sessions DG, Lenox J, Spector GJ, Chao C, Chaudry OA. Analysis of treatment results for base of tongue cancer. Laryngoscope. 2003 Jul;113(7):1252-61. doi: 10.1097/00005537-200307000-00026. PMID 12838028
- [Result] Weinstein GS, O'Malley BW Jr, Magnuson JS, Carroll WR, Olsen KD, Daio L, Moore EJ, Holsinger FC. Transoral robotic surgery: a multicenter study to assess feasibility, safety, and surgical margins. Laryngoscope. 2012 Aug;122(8):1701-7. doi: 10.1002/lary.23294. Epub 2012 Jul 2. PMID 22752997
- [Result] Ibrahim AS, Civantos FJ, Leibowitz JM, Thomas GR, Arnold DJ, Franzmann EJ, Nicolli EA, Lo K, Nemeth Z, Sargi ZB, Weed DT. Meta-analysis comparing outcomes of different transoral surgical modalities in management of oropharyngeal carcinoma. Head Neck. 2019 Jun;41(6):1656-1666. doi: 10.1002/hed.25647. Epub 2019 Jan 28. PMID 30689251
- [Result] Kamran SC, Qureshi MM, Jalisi S, Salama A, Grillone G, Truong MT. Primary surgery versus primary radiation-based treatment for locally advanced oropharyngeal cancer. Laryngoscope. 2018 Jun;128(6):1353-1364. doi: 10.1002/lary.26903. Epub 2017 Oct 8. PMID 28988426
- [Result] O'Connell D, Seikaly H, Murphy R, Fung C, Cooper T, Knox A, Scrimger R, Harris JR. Primary surgery versus chemoradiotherapy for advanced oropharyngeal cancers: a longitudinal population study. J Otolaryngol Head Neck Surg. 2013 Apr 22;42(1):31. doi: 10.1186/1916-0216-42-31. eCollection 2013. PMID 23663568
- [Result] Stelmes JJ, Gregoire V, Poorten VV, Golusinski W, Szewczyk M, Jones T, Ansarin M, Broglie MA, Giger R, Klussmann JP, Evans M, Bourhis J, Leemans CR, Spriano G, Dietz A, Hunter K, Zimmermann F, Tinhofer I, Patterson JM, Quaglini S, Govaerts AS, Fortpied C, Simon C. Organ Preservation and Late Functional Outcome in Oropharyngeal Carcinoma: Rationale of EORTC 1420, the "Best of" Trial. Front Oncol. 2019 Oct 22;9:999. doi: 10.3389/fonc.2019.00999. eCollection 2019. PMID 31696052
- [Result] Boscolo-Rizzo P, Stellin M, Fuson R, Marchiori C, Gava A, Da Mosto MC. Long-term quality of life after treatment for locally advanced oropharyngeal carcinoma: surgery and postoperative radiotherapy versus concurrent chemoradiation. Oral Oncol. 2009 Nov;45(11):953-7. doi: 10.1016/j.oraloncology.2009.06.005. Epub 2009 Aug 8. PMID 19665919
- [Result] Clark JM, Holmes EM, O'Connell DA, Harris J, Seikaly H, Biron VL. Long-term survival and swallowing outcomes in advanced stage oropharyngeal squamous cell carcinomas. Papillomavirus Res. 2019 Jun;7:1-10. doi: 10.1016/j.pvr.2018.09.002. Epub 2018 Sep 26. PMID 30267774
- [Result] Cano ER, Lai SY, Caylakli F, Johnson JT, Ferris RL, Carrau RL, Snyderman CH, Gooding WE, Simenthal AA Jr, Myers EN. Management of squamous cell carcinoma of the base of tongue with chemoradiation and brachytherapy. Head Neck. 2009 Nov;31(11):1431-8. doi: 10.1002/hed.21111. PMID 19405086
- [Result] Agarwal JP, Mallick I, Bhutani R, Ghosh-Laskar S, Gupta T, Budrukkar A, Murthy V, Sengar M, Dinshaw KA. Prognostic factors in oropharyngeal cancer--analysis of 627 cases receiving definitive radiotherapy. Acta Oncol. 2009;48(7):1026-33. doi: 10.1080/02841860902845839. PMID 19363712
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Behera P, Patro BK. Population Based Cancer Registry of India - the Challenges and Opportunities. Asian Pac J Cancer Prev. 2018 Oct 26;19(10):2885-2889. doi: 10.22034/APJCP.2018.19.10.2885. PMID 30362317
- [Result] Robbins KT, Clayman G, Levine PA, Medina J, Sessions R, Shaha A, Som P, Wolf GT; American Head and Neck Society; American Academy of Otolaryngology--Head and Neck Surgery. Neck dissection classification update: revisions proposed by the American Head and Neck Society and the American Academy of Otolaryngology-Head and Neck Surgery. Arch Otolaryngol Head Neck Surg. 2002 Jul;128(7):751-8. doi: 10.1001/archotol.128.7.751. No abstract available. PMID 12117328
- [Result] Koyfman SA, Ismaila N, Crook D, D'Cruz A, Rodriguez CP, Sher DJ, Silbermins D, Sturgis EM, Tsue TT, Weiss J, Yom SS, Holsinger FC. Management of the Neck in Squamous Cell Carcinoma of the Oral Cavity and Oropharynx: ASCO Clinical Practice Guideline. J Clin Oncol. 2019 Jul 10;37(20):1753-1774. doi: 10.1200/JCO.18.01921. Epub 2019 Feb 27. PMID 30811281
- [Result] Mallampati SR, Gatt SP, Gugino LD, Desai SP, Waraksa B, Freiberger D, Liu PL. A clinical sign to predict difficult tracheal intubation: a prospective study. Can Anaesth Soc J. 1985 Jul;32(4):429-34. doi: 10.1007/BF03011357. PMID 4027773
- [Result] Amin MB, Edge S, Greene F, Byrd DR, Brookland RK, Washington MK, et al., editors. AJCC Cancer Staging Manual [Internet]. 8th ed. Springer International Publishing; 2017 [cited 2020 Feb 24].
- [Result] Chen AY, Frankowski R, Bishop-Leone J, Hebert T, Leyk S, Lewin J, Goepfert H. The development and validation of a dysphagia-specific quality-of-life questionnaire for patients with head and neck cancer: the M. D. Anderson dysphagia inventory. Arch Otolaryngol Head Neck Surg. 2001 Jul;127(7):870-6. PMID 11448365
- [Result] Bjordal K, de Graeff A, Fayers PM, Hammerlid E, van Pottelsberghe C, Curran D, Ahlner-Elmqvist M, Maher EJ, Meyza JW, Bredart A, Soderholm AL, Arraras JJ, Feine JS, Abendstein H, Morton RP, Pignon T, Huguenin P, Bottomly A, Kaasa S. A 12 country field study of the EORTC QLQ-C30 (version 3.0) and the head and neck cancer specific module (EORTC QLQ-H&N35) in head and neck patients. EORTC Quality of Life Group. Eur J Cancer. 2000 Sep;36(14):1796-807. doi: 10.1016/s0959-8049(00)00186-6. PMID 10974628
- [Result] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Result] Martin-Harris B, Brodsky MB, Michel Y, Castell DO, Schleicher M, Sandidge J, Maxwell R, Blair J. MBS measurement tool for swallow impairment--MBSImp: establishing a standard. Dysphagia. 2008 Dec;23(4):392-405. doi: 10.1007/s00455-008-9185-9. Epub 2008 Oct 15. PMID 18855050
- [Result] Noronha V, Patil VM, Joshi A, Mahimkar M, Patel U, Pandey MK, Chandrasekharan A, Dsouza H, Bhattacharjee A, Mahajan A, Sabale N, Agarwal JP, Ghosh-Laskar S, Budrukkar A, D'Cruz AK, Chaturvedi P, Pai PS, Chaukar D, Nair S, Thiagarajan S, Banavali S, Prabhash K. Nimotuzumab-cisplatin-radiation versus cisplatin-radiation in HPV negative oropharyngeal cancer. Oncotarget. 2020 Jan 28;11(4):399-408. doi: 10.18632/oncotarget.27443. eCollection 2020 Jan 28. PMID 32064043
- [Result] Hunsberger S, Zhao Y, Simon R. A comparison of phase II study strategies. Clin Cancer Res. 2009 Oct 1;15(19):5950-5. doi: 10.1158/1078-0432.CCR-08-3205. Epub 2009 Sep 29. PMID 19789306
- See also: Amin MB, Edge S, Greene F, Byrd DR, Brookland RK, Washington MK, et al., editors. AJCC Cancer Staging Manual [Internet]. 8th ed. Springer International Publishing; 2017 [cited 2020 Feb 24]. — https://www.springer.com/gp/book/9783319406176
- See also: Radiation Therapy and Cisplatin With or Without Surgery in Treating Patients With Stage III-IV Oropharyngeal Cancer - Full Text View - ClinicalTrials.gov [Internet]. [cited 2020 Feb 24]. — https://clinicaltrials.gov/ct2/show/NCT01953952
- See also: Doyle DJ, Garmon EH. American Society of Anesthesiologists Classification (ASA Class). In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2020 [ — http://www.ncbi.nlm.nih.gov/books/NBK441940/